CLINICAL TRIAL: NCT04415138
Title: Prospective Evaluation of Robotic-assisted Mitral Surgery With the daVinci X Surgical System: HUMANITAS Gavazzeni Contribution (Studio Dell'Applicazione Della Chirurgia Robotica Con Robot daVinci X (IS4200) di Ultima Generazione Sulla Valvulopatia Mitralica: Contributo di HUMANITAS Gavazzeni)
Brief Title: Evaluation of Robotic-assisted Mitral Surgery With the daVinci X Surgical System
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Cliniche Humanitas Gavazzeni (Other)
Responsible Party: Principal Investigator, Alfonso Agnino, MD, Director of Robotic and Video-Assisted Cardiac Surgery Division, Cliniche Humanitas Gavazzeni
Other Study IDs: GAV 213/20
Record Dates: First submitted 2020-05-21; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Mitral Regurgitation; Surgery
Keywords: Robotic Surgery; Outcomes; Cost analysis
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Robotic-assisted Group
  Interventions: Device: Robotic-assisted mitral valve repair
- Video-assisted Group

INTERVENTIONS:
Device: Robotic-assisted mitral valve repair — Mitral valve repair using robotic technology (DaVinci X platform)
  Groups: Robotic-assisted Group

SUMMARY:
Robotic assistance allows performance of mitral valve operations with a truly minimally invasive and totally thoracoscopic approach, with significant advantages for patients compared to sternotomy-based surgery. Nonetheless, its diffusion has been limited by: 1) significant learning curve and technical requirements; 2) increased immediate financial costs due to dedicated equipment and materials. The aim of the present study is to perform a prospective data collection and evaluation of the in-hospital and follow-up clinical results of mitral valve repair using the last generation DaVinci X robotic platform. A cost-effectiveness analysis of this approach will be also conducted, under a global healthcare system perspective (including the overall patients' pathway starting from diagnosis of mitral valve disease until the completion of the 1st postoperative year). Since the 'competitor' surgical technique is not represented by sternotomy-based mitral surgery, but instead by minimally invasive, video-assisted mitral surgery, patients operated on using such technique will serve as controls.

DETAILED DESCRIPTION:
In an observational, prospective, case-control investigation, the clinical data of all adult (18 years-old or more) patients undergoing robotic-assisted mitral surgery in the Sponsor hospital during the study period will be collected, including preoperative, intraoperative and early postoperative variables. Patients need to be affected by severe mitral regurgitation due to degenerative lesions and be eligible to robotic-assisted surgery. An informed consent for inclusion in the study and management of personal data will be asked from all participants. A total of 30 Baseline variables, 9 intraoperative variables, 26 early postoperative variables and 55 follow-up variables will be collected. Systematic in-house follow-up (clinical and echocardiographic) will be performed at the 3rd, 6th and 12th postoperative months. The database will be managed by research assistants under the supervision of the surgical team. Operations will be performed according to the Institutional protocol using the DaVinci X robotic platform by a trained multidisciplinary team including cardiac surgeons, anesthesiologists, cardiologists, perfusionists and scrub nurses.

The same data will be obtained for all patients undergoing minimally invasive, video-assisted non-robotic-assisted mitral repair during the study period. These patients will serve as controls.

Study Endpoints will include procedural success, early postoperative complications, postoperative functional recovery (both immediate and at follow-up), echocardiographic results of mitral repair.

Such data will be compared with those from control patients undergoing minimally invasive, non-robotic-assisted mitral surgery in our Department during the study period.

In cooperation with Hospital Administration Team, all direct and indirect costs (Euros) associated with the in-hospital pathway of each individual patient will be quantified (17 variables per patient within a separate database). Data collection will be expanded to any hospitalisation occurring during the 1st postoperative year. Such data collection will include patients undergoing both the robotic-assisted and the minimally invasive video-assisted non-robotic-assisted strategy.

Data will be analysed using intergoup comparison statistical tests.

ELIGIBILITY:
Inclusion Criteria:

* Aged at least 18, willing to complete the study follow-up, having signed the informed consent for participation and data management.
* Severe mitral regurgitation due to degenerative disease with indication to mitral repair surgery.
* If of female gender, being neither pregnant nor lactating.

Exclusion Criteria:

* Previous right chest surgery or severe right intrapleural adhesions.
* Diameter of femoral arteries equal or lesser than 6 mm.
* Left ventricular systolic dysfunction (LVEF <60%).
* Severe right ventricular dysfunction.
* Aortic valve regurgitation >1+/4+.
* Pulmonary artery hypertension (PASP >50 mmHg).
* Chest deformities preventing either robotic-assisted or minimally invasive video-assisted surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by severe mitral regurgitation due to degenerative disease (Leaflet prolapse/flail) with indication to surgical mitral repair using either a robotic-assisted approach or a minimally invasive video-assisted non-robotic-assisted approach. Includes patients referred to a tertiary cardiac surgical centre.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-03-10 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Duration of ICU stay (hours) and Hospital stay (days and hours) | Up to 30 days after index surgery.
  Duration of stay inside healthcare facility providing index operation. Average value and standard deviation will be presented.
Rate of Major Adverse Cerebral and Cardiovascular Events (MACCE) | Day of index surgery until 30th postoperative day or discharge
  Rate of stroke/TIA, myocardial infarction, cardiac reoperation (presented through both individual and aggregated rates).
Economic evaluation (direct and indirect costs). | Up to 90 days after index surgery.
  Direct and indirect costs associated with robotic-assisted mitral surgery. These will be evaluated for each individual patient and expressed in Euros, under the form of average value and standard deviation. Direct costs will be categorized as follows: total supplies, total drugs, unit operating costs, unit supporting costs).

SECONDARY OUTCOMES:
Rate of residual mitral regurgitation (Early). | Up to 60 days after index surgery.
  Data will be obtained from pre-discharge echocardiography. Residual Mitral Regurgitation is defined as being at least of degree 2+/4+ according to current Echocardiography recommendations.
Rate of residual mitral regurgitation (follow-up). | From the 3rd until the 12th month after index surgery.
  Data will be obtained from echocardiography performed at the 3rd, 6th and 12th postoperative months. Residual Mitral Regurgitation is defined as being at least of degree 2+/4+ according to current Echocardiography recommendations.

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniche HUMANITAS Gavazzeni, Bergamo, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Nifong LW, Chitwood WR, Pappas PS, Smith CR, Argenziano M, Starnes VA, Shah PM. Robotic mitral valve surgery: a United States multicenter trial. J Thorac Cardiovasc Surg. 2005 Jun;129(6):1395-404. doi: 10.1016/j.jtcvs.2004.07.050. PMID 15942584
- [Result] Agnino A, Parrinello M, Panisi P, Anselmi A. Novel nonresectional posterior leaflet remodeling approach for minimally invasive mitral repair. J Thorac Cardiovasc Surg. 2017 Oct;154(4):1247-1249. doi: 10.1016/j.jtcvs.2017.04.076. Epub 2017 May 23. No abstract available. PMID 28606395
- [Result] Rodriguez E, Nifong LW, Bonatti J, Casula R, Falk V, Folliguet TA, Kiaii BB, Mack MJ, Mihaljevic T, Smith JM, Suri RM, Bavaria JE, MacGillivray TE, Chitwood WR Jr. Pathway for surgeons and programs to establish and maintain a successful robot-assisted adult cardiac surgery program. J Thorac Cardiovasc Surg. 2016 Jul;152(1):9-13. doi: 10.1016/j.jtcvs.2016.05.018. No abstract available. PMID 27343904
- [Result] Gillinov AM, Mihaljevic T, Javadikasgari H, Suri RM, Mick SL, Navia JL, Desai MY, Bonatti J, Khosravi M, Idrees JJ, Lowry AM, Blackstone EH, Svensson LG. Early results of robotically assisted mitral valve surgery: Analysis of the first 1000 cases. J Thorac Cardiovasc Surg. 2018 Jan;155(1):82-91.e2. doi: 10.1016/j.jtcvs.2017.07.037. Epub 2017 Aug 1. PMID 28893396
- [Result] Hawkins RB, Mehaffey JH, Mullen MG, Nifong WL, Chitwood WR, Katz MR, Quader MA, Kiser AC, Speir AM, Ailawadi G; Investigators for the Virginia Cardiac Services Quality Initiative. A propensity matched analysis of robotic, minimally invasive, and conventional mitral valve surgery. Heart. 2018 Dec;104(23):1970-1975. doi: 10.1136/heartjnl-2018-313129. Epub 2018 Jun 18. PMID 29915143
- [Result] Suri RM, Thompson JE, Burkhart HM, Huebner M, Borah BJ, Li Z, Michelena HI, Visscher SL, Roger VL, Daly RC, Cook DJ, Enriquez-Sarano M, Schaff HV. Improving affordability through innovation in the surgical treatment of mitral valve disease. Mayo Clin Proc. 2013 Oct;88(10):1075-84. doi: 10.1016/j.mayocp.2013.06.022. PMID 24079678
- [Result] Agnino A, Antonazzo A, Albano G, Panisi P, Gerometta P, Piti A, Anselmi A. Strategy-specific durability of mitral valve repair through the video-assisted right minithoracotomy approach. J Cardiovasc Med (Hagerstown). 2019 Mar;20(3):137-144. doi: 10.2459/JCM.0000000000000753. PMID 30601192
- [Result] Agnino A, Graniero A, Roscitano C, Villari N, Marvelli A, Verhoye JP, Anselmi A. Continued follow-up of the free margin running suture technique for mitral repair. Eur J Cardiothorac Surg. 2020 Oct 1;58(4):847-854. doi: 10.1093/ejcts/ezaa122. PMID 32380519